CLINICAL TRIAL: NCT05126251
Title: Efficacy and Safety of Tangningtongluo Tablet in People With Prediabetes : a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Tangningtongluo Tablet for People With Prediabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Shuyu Yang, Researcher, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZY-KJS-2021-006
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — tangningtongluo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangningtongluo group (Experimental): 1. Tangningtongluo tablet will be used in this arm. Patients should take medicine with warm water about 30min after meal. (1.6g/time, twice a day) According to the above usage and dosage, take 12 weeks continuously. After 12 weeks, the researcher decided whether the subjects entered the extended trial according to the wishes of the subjects, and continued to use the drug until 24 weeks.
  2. Lifestyle intervention
  Interventions: Drug: Tangningtongluo tablet; Behavioral: lifestyle intervention
- Placebo group (Placebo Comparator): Placebo of Tangningtongluo tablet will be used in this arm. Patients should take medicine with warm water about 30min after meal. (2.0g/time, twice a day) According to the above usage and dosage, take 12 weeks continuously. After 12 weeks, the researcher decided whether the subjects entered the extended trial according to the wishes of the subjects, and continued to use the drug until 24 weeks.
  2） Lifestyle intervention
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Drug: Tangningtongluo tablet — Tangningtongluo Tablet is an in-hospital preparation of Guizhou bailing. It is used for diabetes caused by deficiency of Qi and Yin. The symptoms include thirst, drinking, overeating, polyuria, weight loss, shortness of breath, fatigue, hand, foot and heart heat and blurred vision; Type 2 diabetes and diabetic retinopathy see the above syndrome. The present study shows that Tangningtongluo Tablet have certain hypoglycemic effects in diabetic animal models and diabetic patients, and may improve insulin sensitivity in diabetic mice.It is speculated that the drug may be effective for prediabetes. (0.4g/tablet,Plate(12 pills/plate ×3 plates/box))
  Arms: Tangningtongluo group
Behavioral: lifestyle intervention — Avoid overeating, avoid large intake of high-calorie, high-fat foods, live a regular life, avoid sitting for a long time, strengthen exercise and reduce weight.

SUMMARY:
Prediabetes is an intermediate transition to hyperglycemia between normal blood glucose and diabetes, including impaired fasting glucose (IFG), impaired glucose tolerance (IGT)and the presence of a combination of the two.

At present, the prediabetes population in China is very large. Timely detection of this sub-health population and effective intervention are the key to prevent or delay diabetes and related complications. Basic research showed that Tangningtongluo had a good hypoglycemic effect on db/db diabetic mice and STZ induced diabetic rats, and could alleviate pancreatic islet destruction and insulin resistance to some extent.

In this study, the therapeutic effects of Tangningtongluo pian provided by Guizhou bailing Enterprise Group Pharmaceutical Co., Ltd on patients with prediabetes was evaluated clinically. A multi-center, randomized, double-blind, placebo-controlled clinical trial was designed to provide evidence-based medical evidence for Tangningtongluo pian in the treatment of prediabetes . In the design of this trial, the therapeutic effects and safety of Tangningtongluo pian in the treatment of prediabetes were evaluated with Tangningtongluo pian in the treatment group and placebo in the control group.

DETAILED DESCRIPTION:
Prediabetes is an intermediate transition to hyperglycemia between normal blood glucose and diabetes, including impaired fasting glucose (IFG), impaired glucose tolerance (IGT)and the presence of a combination of the two.

At present, the prediabetes population in China is very large. Timely detection of this sub-health state and effective intervention are the key to prevent or delay diabetes and related complications. Prediabetes is mainly IGT, and its core pathophysiological basis is insulin resistance. The existing western medicine can improve insulin resistance to varying degrees, but it can not prevent diabetes. Tangning Tongluo is an in-hospital preparation of Guizhou bailing. It is used for diabetes caused by deficiency of Qi and Yin. The symptoms include thirst, drinking, overeating, polyuria, weight loss, shortness of breath, fatigue, hand, foot and heart heat and blurred vision; Type 2 diabetes and diabetic retinopathy see the above syndrome.Basic research showed that Tang Ning Tong Luo had a good hypoglycemic effect on db/db diabetic mice and STZ induced diabetic rats, and could alleviate pancreatic islet destruction and insulin resistance to some extent. In addition, the drug has a certain retarding effect on diabetic nephropathy animal models [renal function, renal pathology, urinary protein (3+ to 2+)] and fundus lesions, and also improves liver function and myocardial enzymes. Further mechanism studies show that Tangning Tongluo exerts its anti-inflammatory, hypoglycemic and obesity induced insulin resistance effects by up regulating the expression of sequence binding protein (SBP) 2 in macrophages ; In addition, mip1 was inhibited γ/ CCR1 axis improves in diabetic retinopathy.It is speculated that the drug may be effective for prediabetes In this study, the therapeutic effects of Tangningtongluo pian provided by Guizhou bailing Enterprise Group Pharmaceutical Co., Ltd on patients with prediabetes was evaluated clinically. A multi-center, randomized, double-blind, placebo-controlled clinical trial was designed to provide evidence-based medical evidence for Tangningtongluo pian in the treatment of prediabetes .

In the design of this trial, the therapeutic effects and safety of Tangningtongluo pian in the treatment of prediabetes were evaluated with Tangningtongluo pian in the treatment group and placebo in the control group.

ELIGIBILITY:
Inclusion Criteria:

* FPG 5.6mmol/L~6.9mmol/L or OGTT 2H blood glucose 7.8mmol/L~11.0mmol/L or HbA1c 5.7%~6.4%, the above 3 indicators need to meet at least 2 items；
* Age 18 ~ 70 years old (including boundary value);
* Patients who voluntarily signed the informed consent and had conditional follow-up.

Exclusion Criteria:

* Regularly take drugs affecting blood glucose within 1 month before screening, such as hypoglycemic drugs, glucocorticoids, niacin β- Adrenergic agonists, thyroid hormones, contraceptives, diazoxide, diuretics, phenytoin sodium γ- Interferon, etc;
* Combined with various diseases that may significantly shorten life expectancy, such as malignant tumors, severe organ failure and so on;
* Combined with various diseases that may seriously affect the subject's participation in the test, such as psychosis, serious motor system abnormalities, etc;
* Combined ALT or ast > 2.5 times the upper limit of normal value, or serum creatinine > 1.5mg/dl;
* Allergic to the test drug or its components;
* Pregnant or lactating women, or women who have pregnancy plans from the study period to 3 months after the last administration, or men who are unwilling to take a medically recognized effective non drug contraceptive measure.
* Chronic diarrhea caused by inflammatory bowel disease and irritable bowel syndrome;
* The investigator believes that it is inappropriate to be included in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity index | Baseline, 12weeks, 24weeks(if necessary)
  The change of Matsuda index value from baseline calculated according to three-point OGTT (0, 30min, 120min).
Pancreatic β-cell function indicators | Baseline, 12weeks, 24weeks(if necessary)
  The change of Pancreatic β-cell function indicators from baseline according to insulin source index and insulin disposal index.
HbA1c | Baseline, 12weeks, 24weeks(if necessary)
  The change of HbA1c from baseline
Metabolic index | Baseline, 12weeks, 24weeks(if necessary)
  Changes of fasting blood glucose, OGTT 2H blood glucose,body weight, BMI, waist circumference, waist hip ratio, blood lipid (TC, TG, HDL-C, LDL-C), free fatty acid and blood uric acid from baseline
Diabetes incidence rate | Baseline, 12weeks, 24weeks(if necessary)
  Diabetes incidence rate of experimental group=Number of people diagnosed with diabetes/The sample size of experimental group Diabetes incidence rate of placebo group=Number of people diagnosed with diabetes/The sample size of placebo group
The rate of blood glucose reversed to normal | Baseline, 12weeks, 24weeks(if necessary)
  The rate of blood glucose reversed to normal in experimental group=Number of people blood glucose reversed to normal/The sample size of experimental group The rate of blood glucose reversed to normal in placebo group=Number of people blood glucose reversed to normal/The sample size of placebo group
Changes in the proportion of subjects diagnosed with fatty liver from baseline | Baseline, 12weeks, 24weeks(if necessary)
  Changes in the proportion of the experimental group=The proportion of subjects diagnosed with fatty liver after treatment in the experimental group-The proportion of subjects diagnosed with fatty liver in the experimental group in baseline； Changes in the proportion of the placebo group=The proportion of subjects diagnosed with fatty liver after treatment in the placebo group-The proportion of subjects diagnosed with fatty liver in the placebo group in baseline；
Vascular endothelial function indexes: PAI-1 | Baseline, 12weeks, 24weeks(if necessary)
  Changes of PAI-1 from baseline
Vascular endothelial function indexes: NO | Baseline, 12weeks, 24weeks(if necessary)
  Changes of NO from baseline
Vascular endothelial function indexes: ET-1 | Baseline, 12weeks, 24weeks(if necessary)
  Changes of ET-1 from baseline
Inflammatory factor index: TNF-α | Baseline, 12weeks, 24weeks(if necessary)
  Changes of TNF-α from baseline
Inflammatory factor index: IL-6 | Baseline, 12weeks, 24weeks(if necessary)
  Changes of IL-6 from baseline
Inflammatory factor index: IL-2 | Baseline, 12weeks, 24weeks(if necessary)
  Changes of IL-2 from baseline
Inflammatory factor index: IL-1β | Baseline, 12weeks, 24weeks(if necessary)
  Changes of IL-1β from baseline
Inflammatory factor index: adiponectin | Baseline, 12weeks, 24weeks(if necessary)
  Changes of adiponectin from baseline
Inflammatory factor index: hsCRP | Baseline, 12weeks, 24weeks(if necessary)
  Changes of hsCRP from baseline
Inflammatory factor index: FGF-21 | Baseline, 12weeks, 24weeks(if necessary)
  Changes of FGF-21 from baseline
Urinary albumin creatinine ratio (UACR) | Baseline, 12weeks, 24weeks(if necessary)
  Changes of Urinary albumin creatinine ratio (UACR) from baseline
Incidence of diabetic retinopathy | Baseline, 12weeks, 24weeks(if necessary)
  Incidence of diabetic retinopathy of experimental group=Number of people diagnosed with diabetic retinopathy/The sample size of experimental group Incidence of diabetic retinopathy of placebo group=Number of people diagnosed with diabetic retinopathy/The sample size of placebo group
Carotid artery intima-media thickness | Baseline, 12weeks, 24weeks(if necessary)
  Changes of Carotid artery intima-media thickness measured by an ultrasound scanner from baseline
The scores of prediabetes symptom questionnaire | Baseline, 12weeks, 24weeks(if necessary)
  Changes of the score of prediabetes symptom questionnaire from baseline . This scale is self-made and includes 15 symptoms. Each symptom scores 0-3 points, and the total score is 45 points. The higher the score, the more severe the symptoms.
The scores of short form health survey (SF-36) | Baseline, 12weeks, 24weeks(if necessary)
  Changes of the MOS 36 item short form health survey (SF-36) scores from baseline，the minimum and maximum values of the survey are 156 and 37 respectively, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided